CLINICAL TRIAL: NCT00001333
Title: Phase I Study of Intrathecal Topotecan
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 930085; 93-C-0085
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-01

CONDITIONS: Leukemia; Lymphoma; Meningeal Neoplasms
Keywords: Intraventricular; Meningeal Malignancy; NSC 609699; SKF 104864; Topoisomerase 1
MeSH Terms: conditions — Leukemia; Lymphoma; Meningeal Neoplasms | interventions — Topotecan

INTERVENTIONS:
Drug: topotecan

SUMMARY:
The purpose of this study is to determine the qualitative and quantitative toxicity of intrathecal topotecan, a topoisomerase I inhibitor, in patients with meningeal malignancies refractory to conventional therapy (radiation therapy and chemotherapy).

DETAILED DESCRIPTION:
The purpose of this study is to determine the qualitative and quantitative toxicity of intrathecal topotecan, a topoisomerase I inhibitor, in patients with meningeal malignancies refractory to conventional therapy (radiation therapy and chemotherapy). A safe dose of topotecan that can be recommended for intrathecal administration in subsequent phase II studies will be established in a limited dosage escalation schedule. The CSF pharmacokinetics of intrathecal topotecan will also be studied. Topotecan will be administered intrathecally on a bi-weekly basis for four to six weeks, followed by weekly administration for 1 month, twice monthly administration for four months and then monthly IT administration.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Leukemia, lymphoma, or solid tumor with overt meningeal involvement considered refractory to conventional therapy.

CSF leukemic cell count at least 5 per cubic millimeter with evidence of blast cells on cytospin or cytology required for leukemia and lymphoma patients.

Tumor cells on cytospin or cytology or measurable meningeal disease on CT or MRI required for patients with solid tumors.

No clinical evidence of obstructive hydrocephalus or compartmentalization of the CSF flow as documented by indium-111- or technetium-99-DPTA flow study.

PRIOR/CONCURRENT THERAPY:

At least 1 week since CNS therapy.

Biologic Therapy: Recovery from toxic effects of prior immunotherapy required.

Chemotherapy:

Recovery from toxic effects of prior chemotherapy required.

No concomitant therapy to treat meningeal malignancy (intrathecal or systemic).

Concomitant chemotherapy to control systemic disease or bulk CNS disease allowed except: Investigational agents. Agents that penetrate the CNS (e.g., high-dose methotrexate, thiotepa, high-dose cytarabine, fluorouracil, intravenous mercaptopurine).

Agents known to have serious unpredictable CNS side effects.

Endocrine Therapy: Not specified.

Radiotherapy: Recovery from toxic effects of prior radiotherapy required. Patient eligible if flow restored following focal radiotherapy to the blockage site.

Surgery: Not specified.

PATIENT CHARACTERISTICS:

Age: 3 and over (older patients giving consent will be enrolled before the very young, if possible).

Performance status: ECOG 0-2.

Life expectancy: At least 8 weeks.

Hematopoietic: See Disease Characteristics.

Hepatic: Bilirubin less than 2.0 mg/dL, SGPT less than 3 times normal.

Renal: Creatinine less than 1.5 mg/dL.

Metabolic: Serum electrolytes (including calcium and phosphate) normal.

Other: No significant systemic illness (e.g., infection). Not pregnant or lactating.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 1993-02; Study Completion 2000-12

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Rowinsky EK, Grochow LB, Hendricks CB, Ettinger DS, Forastiere AA, Hurowitz LA, McGuire WP, Sartorius SE, Lubejko BG, Kaufmann SH, et al. Phase I and pharmacologic study of topotecan: a novel topoisomerase I inhibitor. J Clin Oncol. 1992 Apr;10(4):647-56. doi: 10.1200/JCO.1992.10.4.647. PMID 1312588
- [Background] Adamson PC, Balis FM, Arndt CA, Holcenberg JS, Narang PK, Murphy RF, Gillespie AJ, Poplack DG. Intrathecal 6-mercaptopurine: preclinical pharmacology, phase I/II trial, and pharmacokinetic study. Cancer Res. 1991 Nov 15;51(22):6079-83. PMID 1933871
- [Background] Blaney SM, Balis FM, Cole DE, Craig C, Reid JM, Ames MM, Krailo M, Reaman G, Hammond D, Poplack DG. Pediatric phase I trial and pharmacokinetic study of topotecan administered as a 24-hour continuous infusion. Cancer Res. 1993 Mar 1;53(5):1032-6. PMID 8439950